CLINICAL TRIAL: NCT06833138
Title: Atrioventricular (AV) Node Ablation and Conduction System Pacing in Patients With Well Controlled Permanent Atrial Fibrillation (AF), Heart Failure and Preserved Ejection Fraction: Heart Rate Regularization vs. Medical Rate Control
Brief Title: Atrioventricular Node Ablation and Conduction System Pacing in Patients With Well Controlled Permanent Atrial Fibrillation (AF), Heart Failure and Preserved Ejection Fraction: Heart Rate Regularization Versus Medical Rate Control
Acronym: HF-RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Medtronic France SAS (Industry); ClinSearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Atrial Fibrillation, Persistent
Keywords: Heart failure; Cardiac Resynchronization Therapy; Conduction System Pacing
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 Intervention arm: Conduction system pacing (pacemaker implantation) + atrioventricular node ablation Control arm: optimal pharmacological therapy
Who Masked: Outcomes Assessor
Masking Description: Clinical outcomes will be adjudicated by the investigator and reviewed by the Clinical Events Committee, which will be blinded to treatment received by the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group with pacemaker implantation and atrioventricular node ablation (Experimental): Pacemaker implantation and atrioventricular node ablation will be performed within a one week period after the randomization.Pharmacological heart failure therapy will be optimized according to current guidelines.
  Interventions: Procedure: pacemaker implantation; Procedure: atrioventricular node ablation; Device: Pacemaker programming
- Control (No Intervention): Conventional care support. The rate control therapy will be optimized to achieve a resting heart rate of <110 beats per minute. Pharmacological heart failure therapy will be optimized according to current guidelines.

INTERVENTIONS:
Procedure: pacemaker implantation — The Medtronic 3830 lead should be used as the Conduction System Pacing lead. However, in case of unsuccessful implantation with the 3830 lead, a stylet-driven lead can be used as an alternative.
  Arms: Intervention group with pacemaker implantation and atrioventricular node ablation
Procedure: atrioventricular node ablation — Right-sided atrioventricular junction ablation will be attempted first with a radiofrequency catheter. The choice of the catheter will be at the discretion of the physician. The catheter will be advanced to the His Bundle and then slightly withdrawn proximally and caudally in order to target the compact atrioventricular node. Repeated ablation procedures will be recommended during follow-up if regression of atrioventricular block occurs.
  Arms: Intervention group with pacemaker implantation and atrioventricular node ablation
Device: Pacemaker programming — The pacemaker device will be programmed in VVIR mode at a lower rate of 75 beats per minute in bipolar mode for sensing and pacing
  Arms: Intervention group with pacemaker implantation and atrioventricular node ablation

SUMMARY:
The goal of this clinical trial is to assess the clinical efficacy of physiological pacing combined with atrioventricular node ablation, in patients with Heart Failure with preserved Ejection Fraction (HFpEF) and well controlled permanent atrial fibrillation.The main question it aims to answer is that heart rate regularization added to physiological pacing - preventing the deleterious effect of right ventricular apical pacing - would reduce mortality and heart failure hospitalizations.

Researchers will compare physiological pacing combined with atrioventricular node ablation (intervention arm) versus optimal pharmacological therapy (control arm) to see if physiological pacing combined with atrioventricular node ablation reduce time to the composite of all-cause mortality or hospitalization due to heart failure or intravenous diuretics (time frame 24 months).

Participants will :

* Be randomized in intervention arm or control arm.
* Visit the clinic 3 months, 12 months and 24 months after the randomization for checkups and tests.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction is a major public health issue affecting 4.9% of general population aged ≥ 60 years. It accounts for more than half of all heart failure hospital admissions. Atrial fibrillation is very common in this diseased population as pathophysiologies are highly interrelated. Atrial fibrillation occurs in two thirds of Heart failure with preserved ejection patients at some point in the natural history and confers a poor prognosis. Therapeutic alternatives are currently limited as patients with permanent Atrial fibrillation and Heart failure with preserved ejection are often treated with drug therapies for lenient rate control.

Recently, the APAF-CRT mortality trial demonstrated a reduction in mortality and hospitalization in Heart Failure and Atrial fibrillation patients treated with Atrioventricular node ablation plus Cardiac Resynchronization Therapy versus pharmacological rate control, irrespective of their baseline Ejection Fraction. The optimal rate regularization achieved with atrioventricular node ablation emerges as the main determinant of reduction in mortality and hospitalization. This conclusion is supported by old robust physiology studies showing that beat-to-beat heart rate irregularity has significant hemodynamic effects and notably decreases cardiac output. However, no specific trials have been conducted in patients with Heart failure with preserved ejection, a population for whom treatment strategies that effectively improve outcomes are sparse. We aim at analyzing the benefit of heart rate regularization and physiological pacing in patients with Heart failure with preserved ejection (Left Ventricular Ejection Fraction ≥ 50%) and permanent Atrial Fibrilation.

We hypothesize that heart rate regularization added to physiological pacing - preventing the deleterious effect of right ventricular apical pacing - would reduce mortality and Heart Failure hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial fibrilation > 6 months
* Preserved Left Ventricular Ejection Fraction ≥ 50%
* ≥ 1 heart failure hospitalization in the previous year
* NYHA (New York Heart Association) score ≥ 2
* Presence of at least one of the following criteria related to diastolic dysfunction:

  * E/e' ratio > 9
  * Left Ventricular mass > 95 g/m2 (female) or > 115 g/m2 (male) with h/R ratio > 0.42
  * NT pro BNP (B-type Natriuretic Peptide) > 365 pg/mL or BNP (B-type Natriuretic Peptide) > 105 pg/mL
* Narrow QRS ≤ 120 ms
* Average heart rate ≤ 110/min on 24 hours Holter monitoring
* Age over 18-year-old
* Capacity to understand the nature of the study, legal ability and willingness to give informed consent
* Patient covered by a social insurance
* Effective contraception and a negative pregnancy test in women of a childbearing age

Exclusion Criteria:

* Patient eligible for atrial fibrilation catheter ablation
* Life expectancy < 12 months
* Severe chronic kidney disease (estimated Glomerular Filtration Rate ≤ 20 ml/1,73 m2)
* Severe respiratory disease (severe chronic obstructive pulmonary disease with Gold ≥ 3 and/or chronic oxygen therapy)
* Class III obesity (Body Mass Index ≥ 40)
* Confirmed or suspected infiltrative cardiomyopathy (amyloidosis, sarcoidosis, Fabry disease, others)
* Obstructive hypertrophic cardiomyopathy
* Previous implanted devices (Pacemaker / Implantable Cardioverter-Defibrillator / Cardiac Resynchronization Therapy)
* Other indication for pacemaker implantation
* Indication for implantable cardioverter-defibrillator
* Ambulatory ≤ 50% of time
* Pregnant women
* Breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to the composite of all-cause mortality or hospitalization due to heart failure or intravenous diuretics. | 24 months
  Delay between randomization and death or hospitalization or intravenous diuretics due to heart failure

SECONDARY OUTCOMES:
Time to all-cause mortality | 24 months
  Delay between randomization and death (all-cause).
Time to Cardiovascular mortality | 24 months
  Delay between randomization and death due to cardiovascular disease.
Time to heart failure hospitalization | 24 months
  Delay between randomization and hospitalization due to heart failure.
Change in New York Heart Association score | 24 months
  Evolution of the functional status measured by New York Heart Association score between randomization and 24 months follow up visit. From II (mild), III (moderate) to IV (severe).
Change in B-type natriuretic peptide level | 24 months
  Evolution of B-type natriuretic peptide (BNP) level between randomization and 24 months follow up visit.
Major adverse events following pacemaker implantation | 24 months
  Record of safety information about pacemaker implantation procedure
Major adverse events following atrioventricular node ablation | 24 months
  Record of safety information about atrioventricular node ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ANSELME, MD, Principal Investigator — CHU de Rouen, France; Corentin CHAUMONT, MD, Study Director — CHU de Rouen, France
Locations (15):
- Belgium (3):
  - OLV Aalst, Aalst
  - UZ Leuven, Leuven
  - Clinique St Pierre Ottignies, Ottignies-Louvain-la-Neuve
- France (12):
  - CHRU de Brest - Hôpital de la Cavale Blanche, Brest
  - CHRU de Caen, Caen
  - CHRU de Tours - Trousseau, Chambray-lès-Tours
  - CHU Grenoble Alpes, Grenoble
  - Groupe Hospitalier La Rochelle-Ré-Aunis, La Rochelle
  - CHRU Lille, Lille
  - GHICL Allome - Hôpital St Philibert, Lomme
  - Clinique Millenaire, Montpellier
  - CHU de Nantes - Hôpital Nord Laennec, Nantes
  - CHU de Bordeaux - Hôpital Cardiologique du Haut-Lévèque, Pessac
  - CHU Poitiers, Poitiers
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No